CLINICAL TRIAL: NCT07388888
Title: Comparative Evaluation of Anti-Bacterial Efficacy Of Two Different Intracanal-Medicaments and Their Effect On Post-Operative Pain Level (A Randomized Clinical Trial)
Brief Title: Antibacterial Effect of Two Different Intracanal Medicaments and Their Effect on Post-operative Pain
Acronym: Ca(OH)2 - CNPs
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana mohamed mustafa nagdy, Dentist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IM012482
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Pulp Necrosis
Keywords: effect of two intracanal medicaments on bacterial load and post operative pain level in mature teeth with necrotic pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- calcium hydroxide (Ca(OH)2) (Active Comparator): intracanal medicament in infected root canal
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)
- Chitosan nano particles (CNPs) (Experimental): intracanal medication in infected root canal
  Interventions: Drug: chitosan nanoparticles gel
- control (No Intervention)

INTERVENTIONS:
Drug: Calcium Hydroxide (Ca(OH)2) — Non setting calcium hydroxide intracanal medicament is injected through the root canal for two weeks
  Arms: calcium hydroxide (Ca(OH)2)
Drug: chitosan nanoparticles gel — Nano chitosan gel is injected through the root canal as an intracanal medicament for two weeks
  Arms: Chitosan nano particles (CNPs)

SUMMARY:
Evaluation of antibacterial effect of two different intracanal medicaments on bacterial load in infected mature permanent teeth and their effect on post-operative pain level.

DETAILED DESCRIPTION:
Microorganisms within the root canal system exist as complex, multispecies biofilms made up of microcolonies that adhere permanently to each other and to surfaces such as dentin. The characteristics of these biofilms-including their composition, thickness, and location-vary according to environmental conditions like nutrient availability, pH, oxygen levels, and exposure to the oral cavity. Endodontic treatment aims to save teeth with damaged pulp tissue, as maintaining natural teeth is essential for proper oral function and overall health. Understanding the specific microorganisms involved in endodontic infections is crucial for explaining disease progression and selecting the most effective treatment strategies.

Because of the intricate anatomy of the root canal system, both mechanical instrumentation and chemical irrigation are required to reduce microbial load. However, chemo-mechanical debridement alone is often insufficient, allowing some bacteria to persist within the canal. As a result, antimicrobial intracanal medicaments have been introduced to enhance disinfection. Although several medicaments are currently used, many show limitations such as microbial resistance or an inability to simultaneously control intracanal infection and periapical inflammation. Additionally, antimicrobial agents may interact with the immune system, potentially suppressing or stimulating immune responses.

Enterococci, particularly *Enterococcus faecalis*, are frequently associated with persistent endodontic infections due to their resistance to treatment and ability to survive harsh conditions. Calcium hydroxide, a material introduced to dentistry in the early 20th century, is widely used as an intracanal medicament but has limited effectiveness against certain bacteria such as *E. faecalis*. Recent interest has focused on nanoparticles, which range from 1 to 100 nm in size and possess unique antimicrobial properties with reduced resistance. Among these, chitosan nanoparticles-derived from chitin found in crustacean exoskeletons-have gained attention for their biocompatibility and antibacterial effects. Effective intracanal medicaments are also important in reducing postoperative pain, which is commonly linked to bacterial irritation following endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* free medical history,
* mature infected permanent single rooted teeth diagnosed clinically and radiographically with adequate coronal structure for proper isolation, temporization and restoration.

Exclusion Criteria:

* Patients who are not included in the age range of the study or having a systemic condition.
* Teeth with severe fractures or resorption or periodontally compromised.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Bacterial load. | two weeks
  Samples will be collected from the infected root canal before and after injection of intracanal medicaments then bacterial colonies will be counted for colony forming units per milliliter (CFU/ml) to assess the effect of the intracanal medicaments used.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) to measure post operative pain level. | 12 hours, 24 hours, 48 hours, 72 hours.
  the patient is given a 10 cm sheet to mark their pain level where (0) represents no pain and (10) the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No